CLINICAL TRIAL: NCT04041375
Title: Using Peer Navigators to Increase Access to VA and Community Resources for Veterans With Diabetes-related Distress
Brief Title: Veteran Support and Resources for Diabetes
Acronym: iNSPiRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 17-221
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Diabetes
Keywords: peer support; mental health; diabetes self-management; community-based participatory research
MeSH Terms: conditions — Diabetes Mellitus; Psychological Well-Being | interventions — Inhalation; Health Resources

STUDY DESIGN:
Intervention Model Description: This is a single-blind, parallel group, randomized trial of a 3-month peer-navigation intervention for Veterans with DM and elevated levels of diabetes-related distress. Participants will be assigned at random (see below) to the intervention (peer navigation with follow-up) or usual care (print materials and encouragement to continue follow-up with health care providers). Assessment of primary, secondary and intermediate end points will occur pre-intervention at baseline and post-intervention at 3 and 6 months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iNSPiRED (Experimental): Peer coaching intervention
  Interventions: Behavioral: iNSPiRED
- Usual Care (Active Comparator): Directory of resources and encouragement to follow-up with Primary Care Physician
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: iNSPiRED — The peer intervention will include approximately 5 to 6 contacts over a 3-month period. Peer navigators are responsible for providing emotional and social support, normalizing the difficulty of living with DM, modeling help-seeking behaviors, and connecting patients with VHA and/or CBOs to address mental health and DM self-management needs. Peer coaches are not responsible for health education directly; rather, they encourage patients to use appropriate programs in which mental health and DM self-management services are provided.
  Other Names: Veteran Support and Resources for Diabetes
  Arms: iNSPiRED
Other: Usual Care — Veterans randomized to the usual care condition will be encouraged to follow-up with their primary care provider and/or specialty providers for management of their health conditions. They will also receive a packet of printed information that includes a list of self-management support resources in the VHA and the local community. They will receive no further specific recommendations
  Arms: Usual Care

SUMMARY:
Patients with diabetes are often challenged by the routine of managing their diabetes, and may experience both stress and medical problems. Diabetes-related medical problems and stress often happen together and affect peoples' ability to live a full, happy and healthy life. Because of this, programs that help with medical problems and stress by teaching ways to better manage diabetes and stress may improve the lives of those with diabetes.

Many excellent programs are available in the VA and in the community that help persons with diabetes better manage their medical problems and stress, but often times Veterans have trouble finding these programs.

The purpose of the study is to see if a telephone-based coaching program improves the physical and emotional health of Veterans with diabetes more than use of a directory of community and VA resources and no coaching. The Veterans who receive the directory of community and VA resources will be given this at the beginning of the study and will access resources as they see fit. Those in the coaching program will be coached by a Veteran with knowledge of diabetes, mental health and community resources who will help them connect to care in the VA and/or community depending on their preference. Examples of resources available in the VA and community include mental health care and programs to help with diet, exercise and learning about how to better manage diabetes.

Veterans who are interested in participating and pass screening will be enrolled in the study for about 6 months. Each enrolled Veteran will have a 50% chance of being enrolled in the coaching group and a 50% chance of being enrolled in the directory group (like the flip of a coin). Both groups will be asked to complete several questionnaires about their health and well-being by telephone. This will occur at the beginning of the study and three and six months later. The questionnaires will take about an hour to complete each time.

DETAILED DESCRIPTION:
Diabetes-related distress, the negative emotional impact of living with diabetes (DM), is a powerful predictor of psychosocial functioning, treatment adherence, and glycemic control. Practice guidelines and consensus statements call for innovative approaches to address DM-related distress. Despite availability of self-management and psychosocial interventions to reduce DM related distress, these interventions are underutilized due to constraints in time, finances, motivation, and resource-awareness. Interventions that leverage traditional medical care and community-based health promotion programs (e.g., DM self-management education (DSME) programs) may enhance the ability of Veterans with DM to engage with a broad and accessible range of resources. Ensuring that Veterans with DM receive adequate self-care support requires interventions that (1) attend to both medical care and diabetes-related distress and (2) improve Veterans' access and engagement with DSME and traditional medical/mental care. Integrating VA and community health services and DSME resources is innovative and affords great opportunities to enhance Veteran outcomes and build VA community partnerships. Engagement of Veterans and community organizations in developing and delivering care responds to the 2016 HSR&D high-priority domain of Health Care Systems Change and aligns with the 2017 VA Under Secretary's priorities of Greater Choice (offering community and VA resources), Efficiency (community and VA coordination), and Timeliness (telephone delivery).

This community-VA partnership and three-month Veteran peer coaching intervention (iNSPiRED) aims to enhance psychological well-being and diabetes self-management behavior in Veterans with DM by facilitating access to and use of healthcare and health promotion resources. The intervention focuses on reducing cognitive and practical barriers to use of services by engaging Veteran peers as coaches and navigators, and by encouraging engagement in health promotion and healthcare services in the VA and the greater community. A secondary goal, integral to the main goal, is to strengthen and integrate VHA partnerships with community-based organizations and Veteran Support Organizations (VSO's).

This is a single-blind, parallel group randomized trial of a 3-month peer navigation intervention for Veterans with DM and elevated levels of DM-related distress. The investigators will recruit Veterans with DM-related distress through existing help-seeking channels within and outside of the VA in partnership with community agencies, VSO's, and the Houston VAMC. Eligible Veterans will be assigned at random to the iNSPiRED intervention (peer navigation and coaching) versus usual care (written resource materials and encouragement to continue follow-up with healthcare providers). Consistent with the focus on the overall emotional impact of DM, the PRIMARY OUTCOME is DM-related distress (DM Distress Scale). In previous studies the DDS has shown strong relationships with psychological symptoms, self-management behaviors, and objective measures of glycemic control. SECONDARY OUTCOMES include anxiety symptoms (Generalized Anxiety Disorder Scale), depression symptoms (Patient Health Questionnaire-8), DM self-management behaviors (DM Self-Management Scale), and self-reported use and new use of VA or community resources. In addition to participant-level outcomes, the investigators will also assess STAKEHOLDER OUTCOMES through a mixed methods process evaluation. The objective will be to measure the impact of stakeholder engagement activities on development and sustainability of VA-community partnerships, trust and communication, and capacity building. Assessment of primary and secondary endpoints will occur at baseline, post-intervention, and at 6 months.

If this project meets intended goals, the investigators will partner with VHA Office of Community Engagement and VHA Specialty Care to implement the intervention for DM and other chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Diagnosis of type 2 DM, per self-report
* Moderate diabetes-related distress (Diabetes Distress Scale [DDS2] mean score of 3 or greater)

Exclusion Criteria:

* Lack of reliable access to a telephone
* Cognitive, sensory, or other impairment that prevents use of a telephone
* Current participation in another diabetes-related counseling or self-management program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Kunik, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications from this research will be made available to the public in electronic form. The investigators will provide a de-identified, quantitative dataset compliant with VA data security policy to the public upon request to the principal investigator. Qualitative data cannot be shared because it has identifiable, sensitive information that cannot be practicably de-identified. Notices advising the public of the availability of the dataset will appear in all publications authored by our research team.
Time Frame: After the data is analyzed and published

REFERENCES:
- [Background] Cully JA, Hundt NE, Fletcher T, Sansgiry S, Zeno D, Kauth MR, Kunik ME, Sorocco K. Brief Cognitive-Behavioral Therapy for Depression in Community Clinics: A Hybrid Effectiveness-Implementation Trial. Psychiatr Serv. 2024 Mar 1;75(3):237-245. doi: 10.1176/appi.ps.20220582. Epub 2023 Sep 7. PMID 37674395
- [Background] Dawson DB, Mohankumar R, Puran D, Nevedal A, Maguen S, Timko C, Kunik ME, Breland JY. Weight Management Treatment Representations: A Novel Use of the Common Sense Model. J Clin Psychol Med Settings. 2023 Dec;30(4):884-892. doi: 10.1007/s10880-023-09946-4. Epub 2023 Feb 24. PMID 36828990
- [Background] Chen GJ, Kunik ME, Marti CN, Choi NG. Cost-effectiveness of Tele-delivered behavioral activation by Lay counselors for homebound older adults with depression. BMC Psychiatry. 2022 Oct 17;22(1):648. doi: 10.1186/s12888-022-04272-9. PMID 36253766
- [Background] Mishra RK, Park C, Momin AS, Rafaei NE, Kunik M, York MK, Najafi B. Care4AD: A Technology-Driven Platform for Care Coordination and Management: Acceptability Study in Dementia. Gerontology. 2023;69(2):227-238. doi: 10.1159/000526219. Epub 2022 Sep 12. PMID 36096091
- [Background] Boykin DM, Wray LO, Funderburk JS, Holliday S, Kunik ME, Kauth MR, Fletcher TL, Mignogna J, Roberson RB 3rd, Cully JA. Leveraging the ExpandNet framework and operational partnerships to scale-up brief Cognitive Behavioral Therapy in VA primary care clinics. J Clin Transl Sci. 2022 Jul 20;6(1):e95. doi: 10.1017/cts.2022.430. eCollection 2022. PMID 36003211
- [Background] Choi NG, Choi BY, Marti CN, Kunik ME. Depression/anxiety symptoms and self-reported difficulty managing medication regimen among community-dwelling older adults. Gen Hosp Psychiatry. 2022 Sep-Oct;78:50-57. doi: 10.1016/j.genhosppsych.2022.07.005. Epub 2022 Jul 15. PMID 35853418

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1,614 Veterans considered for study entry (1,499 referred from VA sources, 110 referred from community sources, 5 referred from both VA and community sources), 1,109 were contacted, 503 were screened, and 219 were eligible/provided informed consent for study participation.
Pre-assignment Details: One participant who provided informed consent withdrew prior to completing baseline/randomization.
Period: Intervention Phase
Arm/Group | iNSPiRED | Usual Care
Started | 110 | 108
Completed | 108 | 106
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Follow-up Phase
Arm/Group | iNSPiRED | Usual Care
Started | 108 | 106
Completed | 101 | 105
Not Completed | 7 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Too ill | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iNSPiRED | Usual Care | Total
Number analyzed (Participants) | 110 | 108 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 59 | 116
  >=65 years | 53 | 49 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.35 (10.31) | 62.37 (11.13) | 62.86 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 98 | 95 | 193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 57 | 59 | 116
  Race: White | 25 | 31 | 56
  Race: Hispanic | 22 | 13 | 35
  Race: Other | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110 | 108 | 218
Education [Count of Participants; unit: Participants]
  High School/GED/No Diploma | 35 | 30 | 65
  Some College or Technical School | 46 | 50 | 96
  Bachelors Degree | 21 | 17 | 38
  Graduate or Professional Degree | 8 | 11 | 19
Annual Income [Count of Participants; unit: Participants]
  <$20k | 41 | 40 | 81
  $20k-$39,999k | 29 | 24 | 53
  $40k-$59,999k | 23 | 22 | 45
  $60k + | 17 | 22 | 39
17-item Diabetes Distress Scale (DDS17)--Total Score [Mean (Standard Deviation); unit: units on a scale] — The content of the DDS17 was developed with the input of people with DM and clinicians with expertise in DM. Items are grouped into 4 subscales: Emotional Burden, Physician-related Distress, Regimen-related Distress, and Interpersonal Distress. Items are rated on a Likert scale indicating the extent to which each factor is distressing. The instrument is scored by computing the average value across items to obtain a total score. Minimum score 1. Maximum score 6. Higher scores indicate worse distress.
  units on a scale | 3.04 (1.11) | 3.06 (1.07) | 3.05 (1.08)
Uses any diabetes medication [Count of Participants; unit: Participants]
  Yes | 107 | 106 | 213
  No | 3 | 2 | 5
Uses insulin [Count of Participants; unit: Participants]
  Yes | 56 | 49 | 105
  No | 54 | 59 | 113
Ever hospitalized for diabetes [Count of Participants; unit: Participants]
  Yes | 27 | 26 | 53
  No | 83 | 82 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change in Diabetes Distress Screening Scale (DDS17)
Description: The content of the DDS17 was developed with the input of people with DM and clinicians with expertise in DM. Items are grouped into 4 subscales: Emotional Burden ("Feeling angry, scared and/or depressed when I think about living with diabetes"), Physician-related Distress ("Feeling that my doctor doesn't take my concerns seriously enough"), Regimen-related Distress ("Not feeling confident in my day-to-day ability to manage diabetes"), and Interpersonal Distress ("Feeling that friends or family don't give me the emotional support that I would like"). Items are rated on a Likert scale indicating the extent to which each factor is distressing, from 1 (no problem) to 6 (a serious problem). The instrument is scored by computing the average value across items to obtain a total score and four subscale scores. Minimum score 1. Maximum score 6. Higher scores indicate worse distress.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
score on a scale
  Baseline--Total Score | 3.0 (1.1) | 3.1 (1.1)
  Baseline--Emotional Burden Subscale | 3.3 (1.3) | 3.3 (1.2)
  Baseline--Physician-Related Distress Subscale | 2.7 (1.3) | 2.6 (1.3)
  Baseline--Regimen-Related Distress Subscale | 3.5 (1.3) | 3.5 (1.2)
  Baseline--Interpersonal Distress Subscale | 2.4 (1.4) | 2.6 (1.5)
  Month 3--Total Score: number analyzed (Participants) | 102 | 103
  Month 3--Total Score | 2.6 (1.1) | 2.4 (1.4)
  Month 3--Emotional Burden Subscale: number analyzed (Participants) | 102 | 103
  Month 3--Emotional Burden Subscale | 2.7 (1.2) | 2.8 (1.1)
  Month 3--Physician-Related Distress Subscale: number analyzed (Participants) | 102 | 103
  Month 3--Physician-Related Distress Subscale | 2.4 (1.2) | 2.4 (1.2)
  Month 3--Regimen-Related Distress Subscale: number analyzed (Participants) | 102 | 103
  Month 3--Regimen-Related Distress Subscale | 2.8 (1.2) | 3.0 (1.2)
  Month 3--Interpersonal Distress Subscale: number analyzed (Participants) | 102 | 103
  Month 3--Interpersonal Distress Subscale | 2.3 (1.4) | 2.2 (1.3)
  Month 6--Total Score: number analyzed (Participants) | 101 | 105
  Month 6--Total Score | 2.6 (1.0) | 2.6 (1.0)
  Month 6--Emotional Burden: number analyzed (Participants) | 101 | 105
  Month 6--Emotional Burden | 2.7 (1.2) | 2.7 (1.1)
  Month 6--Physician-Related: number analyzed (Participants) | 101 | 105
  Month 6--Physician-Related | 2.4 (1.1) | 2.4 (1.2)
  Month 6--Regimen-Related: number analyzed (Participants) | 101 | 105
  Month 6--Regimen-Related | 2.8 (1.1) | 2.9 (1.2)
  Month 6--Interpersonal: number analyzed (Participants) | 101 | 105
  Month 6--Interpersonal | 2.4 (1.4) | 2.2 (1.3)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Total Score - Treatment Effect - Month 3; Test type: Superiority — Treatment effect was modeled via multilevel linear regression with random intercepts for participants. Outcome was regressed on dummy coded categorical indicators of study arm (usual care reference), time point (baseline reference), and arm x time point interaction. Test of the arm x time interaction terms were used to assess treatment effects at months 3 and 6. Models conditioned on race, education, and income as specified a priori; p = 0.42, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.09
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Emotional Burden Subscale - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.32, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.13
Statistical Analysis 3: Comparison: iNSPiRED vs Usual Care; Physician-Related Distress Subscale - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.36, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.13
Statistical Analysis 4: Comparison: iNSPiRED vs Usual Care; Regimen-Related Distress Subscale - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.23, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.17
Statistical Analysis 5: Comparison: iNSPiRED vs Usual Care; Interpersonal Distress Subscale - Treatment Effect - Month 3; Test type: Superiority — Treatment effect was modeled via multilevel linear regression model with random intercepts for participants. Outcome was regressed on dummy coded categorical indicators of study arm (usual care reference), time point (baseline reference), and arm x time point interaction. Test of the arm x time interaction terms were used to assess treatment effects at months 3 and 6. Models conditioned on race, education, and income as specified a priori; p = 0.26, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.18
Statistical Analysis 6: Comparison: iNSPiRED vs Usual Care; Total Score - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.95, Mixed Models Analysis — alpha = 0.05; Treatment Effect = 0.007
Statistical Analysis 7: Comparison: iNSPiRED vs Usual Care; Emotional Burden Subscale - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.92, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.01
Statistical Analysis 8: Comparison: iNSPiRED vs Usual Care; Physician-Related Distress Subscale - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.59, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.07
Statistical Analysis 9: Comparison: iNSPiRED vs Usual Care; Regimen-Related Distress Subscale - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.54, Interaction Term — alpha = 0.05; Interaction Term = -0.08
Statistical Analysis 10: Comparison: iNSPiRED vs Usual Care; Interpersonal Distress Subscale - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.30

2. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities Assessment (SDSCA)
Description: The SDSCA measure is a brief self-report questionnaire of diabetes self-management. It assesses the number of days per week in which respondents engage in diabetes health-related behaviors in the areas of general diet, fruits and vegetable intake, fat intake, physical activity, blood-glucose testing, and foot care. and smoking. Minimum score 0. Maximum score 7 (for each area). Higher scores indicate better self care. Smoking in the last week is also assessed as a binary variable (see separate entry).
Time Frame: Baseline, Month 3, Month 6
Population: Full sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
score on a scale
  Baseline--General Diet | 3.3 (2.1) | 3.3 (2.2)
  Baseline--Specific Diet (Fruits and Vegetables) | 2.8 (2.2) | 2.8 (2.4)
  Baseline--Specific Diet (Fat) | 3.7 (2.0) | 3.1 (2.0)
  Baseline--Physical Activity | 2.7 (2.4) | 2.4 (2.3)
  Baseline--Blood Glucose Testing | 3.0 (2.7) | 3.3 (2.7)
  Baseline--Foot Care | 4.0 (2.2) | 3.7 (2.5)
  Month 3--General Diet: number analyzed (Participants) | 102 | 103
  Month 3--General Diet | 4.2 (1.6) | 3.7 (2.1)
  Month 3--Specific Diet (Fruits and Vegetables): number analyzed (Participants) | 102 | 103
  Month 3--Specific Diet (Fruits and Vegetables) | 3.2 (2.2) | 3.1 (2.6)
  Month 3--Specific Diet (Fat): number analyzed (Participants) | 102 | 103
  Month 3--Specific Diet (Fat) | 3.9 (1.9) | 3.8 (2.0)
  Month 3--Physical Activity: number analyzed (Participants) | 102 | 103
  Month 3--Physical Activity | 3.3 (2.2) | 2.7 (2.2)
  Month 3--Blood Glucose Testing: number analyzed (Participants) | 102 | 103
  Month 3--Blood Glucose Testing | 3.5 (2.6) | 3.9 (2.6)
  Month 3--Foot Care: number analyzed (Participants) | 102 | 103
  Month 3--Foot Care | 4.3 (2.2) | 4.1 (2.4)
  Month 6--General Diet: number analyzed (Participants) | 101 | 105
  Month 6--General Diet | 4.0 (1.6) | 3.8 (1.8)
  Month 6--Specific Diet (Fruits and Vegetables): number analyzed (Participants) | 101 | 105
  Month 6--Specific Diet (Fruits and Vegetables) | 3.2 (2.2) | 3.0 (2.2)
  Month 6--Specific Diet (Fat): number analyzed (Participants) | 101 | 105
  Month 6--Specific Diet (Fat) | 4.0 (1.7) | 3.6 (2.0)
  Month 6--Physical Activity: number analyzed (Participants) | 101 | 105
  Month 6--Physical Activity | 3.1 (2.3) | 2.6 (2.0)
  Month 6--Blood Glucose Testing: number analyzed (Participants) | 101 | 105
  Month 6--Blood Glucose Testing | 3.5 (2.6) | 4.0 (2.4)
  Month 6--Foot Care: number analyzed (Participants) | 101 | 105
  Month 6--Foot Care | 4.4 (2.2) | 3.9 (2.4)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; General Diet - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.03, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.58
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Specific Diet (Fruits and Vegetables) - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.83, Mixed Models Analysis; Interaction Term = 0.07
Statistical Analysis 3: Comparison: iNSPiRED vs Usual Care; Specific Diet (Fat) - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.12, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.44
Statistical Analysis 4: Comparison: iNSPiRED vs Usual Care; Physical Activity - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.17, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.39
Statistical Analysis 5: Comparison: iNSPiRED vs Usual Care; Blood Glucose Testing - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.85, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.06
Statistical Analysis 6: Comparison: iNSPiRED vs Usual Care; Foot Care - Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.94, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.02
Statistical Analysis 7: Comparison: iNSPiRED vs Usual Care; General Diet - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.47, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.19
Statistical Analysis 8: Comparison: iNSPiRED vs Usual Care; Specific Diet (Fruits and Vegetables) - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.82, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.08
Statistical Analysis 9: Comparison: iNSPiRED vs Usual Care; Specific Diet (Fat) - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.66, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.13
Statistical Analysis 10: Comparison: iNSPiRED vs Usual Care; Physical Activity - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.38, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.25
Statistical Analysis 11: Comparison: iNSPiRED vs Usual Care; Blood Glucose Testing - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.68, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.12
Statistical Analysis 12: Comparison: iNSPiRED vs Usual Care; Foot Care - Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.40, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.26

3. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities Assessment (SDSCA)--Number of Participants Who Smoked
Description: The SDSCA measure is a brief self-report questionnaire of diabetes self-management. Any smoking in the last week is assessed as a binary variable. Minimum score 0 (did not smoke). Maximum score 1 (smoked). See separate entry for SDSCA items that measure the number of days per week an activity is performed. Reported counts reflect number of participants who indicated smoking in the last week.
Time Frame: Baseline, Month 3, Month 6
Population: Variation in cell sizes due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
Participants
  Yes - Baseline | 23 | 23
  Yes - Month 3: number analyzed (Participants) | 102 | 103
  Yes - Month 3 | 20 | 24
  Yes - Month 6: number analyzed (Participants) | 101 | 105
  Yes - Month 6 | 20 | 23

4. Secondary Outcome: Change in Patient Health Questionnaire-8 (PHQ-8)
Description: The PHQ-8 is an eight-item questionnaire that assesses the frequency of depression and mood-related symptoms (e.g., "Feeling down, depressed, or hopeless," "Trouble falling or staying asleep, or sleeping too much") over the past 2 weeks. Minimum score 0. Maximum score 24. Higher scores indicate worse depression.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
score on a scale
  Baseline | 11.4 (6.8) | 11.8 (6.6)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 9.3 (6.5) | 9.7 (6.1)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 9.6 (6.7) | 9.6 (6.1)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.93, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.06
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.38, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.63

5. Secondary Outcome: Change in Generalized Anxiety Disorder-7 Questionnaire (GAD-7)
Description: The GAD-7 is a 7-item questionnaire developed as a companion to the PHQ-9 to screen for generalized anxiety disorder and other common anxiety disorders. Items assess the frequency of anxiety symptoms (e.g., "Worrying too much about different things," "Feeling afraid as if something awful might happen") over the past 2 weeks. Minimum score 0. Maximum score 21. Higher scores indicate worse anxiety.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
units on a scale
  Baseline | 10.9 (7.0) | 11.4 (6.4)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 9.3 (6.8) | 9.3 (6.7)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 9.6 (6.9) | 9.2 (6.2)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.66, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.32
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.18, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.99

6. Secondary Outcome: Change in Use of Community Resources (no to Yes)
Description: The investigators will record the Veteran's self-report of any use of community-based resources including mental health care and counseling, DM classes, nutrition services, primary care appointments, and other health-related services. Dichotomous. Yes = care in the community. No= no care in the community
Time Frame: Baseline, Month 6
Population: Full sample
Measure: Number; unit: participants
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 101 | 105
participants | 0 | 0

7. Other Pre Specified Outcome: Change in Use of VHA Resources (no to Yes)
Description: The investigators will record the Veteran's self-report of use of VHA resources including mental health care and counseling, DM classes, nutrition services, primary care appointments, and other health-related services. Dichotomous Yes = care in VHA. No= no care in VHA.
Time Frame: Baseline, Month 6
Population: Full sample
Measure: Number; unit: participants
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 101 | 105
participants | 0 | 0

8. Other Pre Specified Outcome: Change in Patient Activation Measure (PAM)
Description: The Patient Activation Measure (PAM) is designed to measure the extent to which patients endorse subjective ability to self-manage their chronic health conditions. Items assess several aspects of self-management, including knowledge (e.g., "I know what each of my prescribed medications do"), skill (e.g., "I have been able to maintain the lifestyle changes for my health that I have made"), and confidence (e.g., "I am confident I can tell my health care provider concerns I have even when he or she does not ask"). Raw scores: Minimum 13. Maximum 52. Scaled scores ("Activation" scores): Minimum 0.0. Maximum 100.0. Higher scores indicate more patient activation.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
score on a scale
  Baseline | 55.2 (14.3) | 53.2 (12.7)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 60.1 (15.6) | 56.5 (12.4)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 59.1 (15.6) | 56.4 (13.5)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.38, Mixed Models Analysis — alpha = 0.05; Interaction Term = 1.45
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.68, Mixed Models Analysis — alpha = 0.05; Interaction Term = 1.64

9. Other Pre Specified Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS)--PROMIS Short Form v1.0 - Self-Efficacy for Managing Emotions 4a
Description: PROMIS Short Form v1.0 - Self-Efficacy for Managing Emotions 4a measures self-efficacy related to managing emotions. Items are rated on a 5-point scale corresponding to the respondent's degree of confidence for managing various problems or functions. Raw scores: Minimum score 4. Maximum score 20. Scaled scores (T-scores with population mean of 50 and a standard deviation of 10): Minimum score 24.82 Maximum score 63.45. Higher scores indicate higher self-efficacy.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample; number analyzed in one or more rows differs from the overall number analyzed due to missing data.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
T-score
  Baseline | 42.9 (4.1) | 43.0 (4.1)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 43.6 (4.5) | 43.7 (4.3)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 43.5 (4.3) | 43.5 (3.9)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.74, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.19
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.62, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.29

10. Other Pre Specified Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS)--PROMIS Short Form v1.0 - Self-Efficacy for Managing Daily Activities 4a
Description: PROMIS Short Form v1.0 - Self-Efficacy for Managing Daily Activities 4a measures self-efficacy related to managing daily activities. Items are rated on a 5-point scale corresponding to the respondent's degree of confidence for managing various problems or functions. Raw scores: Minimum score 4. Maximum score 20. Scaled scores (T-scores with population mean of 50 and a standard deviation of 10): Minimum score 26.02 Maximum score 59.26. Higher scores indicate higher self-efficacy.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample; number analyzed in one or more rows differs from the overall number analyzed due to missing data.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
T-scores
  Baseline | 41.9 (3.2) | 41.3 (2.9)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 42.5 (3.0) | 41.8 (3.2)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 41.9 (3.3) | 41.6 (3.0)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.72, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.16
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.58, Mixed Models Analysis — alpha = 0.05; Interaction Term = -0.24

11. Other Pre Specified Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS)--PROMIS Short Form v1.0 - Self-Efficacy for Managing Social Interactions 4a
Description: PROMIS Short Form v1.0 - Self-Efficacy for Managing Social Interactions 4a measures self-efficacy related to managing social interactions. Items are rated on a 5-point scale corresponding to the respondent's degree of confidence for managing various problems or functions. Raw scores: Minimum score 4. Maximum score 20. Scaled scores (T-scores with population mean of 50 and a standard deviation of 10): Minimum score 23.08 Maximum score 58.19. Higher scores indicate higher self-efficacy.
Time Frame: Baseline, Month 3, Month 6
Population: Full sample; number analyzed in one or more rows differs from the overall number analyzed due to missing data.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | iNSPiRED | Usual Care
Number analyzed (Participants) | 110 | 108
T-scores
  Baseline | 39.3 (3.9) | 39.8 (4.2)
  Month 3: number analyzed (Participants) | 102 | 103
  Month 3 | 40.5 (3.9) | 40.6 (4.2)
  Month 6: number analyzed (Participants) | 101 | 105
  Month 6 | 40.4 (3.5) | 40.2 (4.2)
Statistical Analysis 1: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 3; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.50, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.36
Statistical Analysis 2: Comparison: iNSPiRED vs Usual Care; Treatment Effect - Month 6; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.18, Mixed Models Analysis — alpha = 0.05; Interaction Term = 0.72

12. Other Pre Specified Outcome: Number of Participants Who Completed the PCORI Ways of Engaging-Engagement Activity Tool (WE-ENACT) Researcher Survey
Description: The investigators will measure stakeholder engagement from the researcher's perspective using a modified version of the PCORI WE-ENACT Researcher Survey, completed annually.
  One group of researchers (the primary investigator and three team members) involved in stakeholder engagement completed the survey together at each time point.
  The Outcome Measure Data Table includes the number of participants who completed the survey (1 group of researchers).
Time Frame: Baseline and every 12 months assessed up to month 48
Measure: Count of Participants; unit: Participants
Groups:
- Researchers: A group of four iNSPiRED researchers involved in stakeholder engagement activities (the primary investigator, two co-investigators, and the project coordinator) completed the PCORI Ways of Engaging-Engagement Activity Tool (WE-ENACT) survey annually to evaluate stakeholder engagement efforts from the researcher perspective. The researchers completed one survey as a team each year.
Arm/Group | Researchers
Number analyzed (Participants) | 1
Participants | 1

13. Other Pre Specified Outcome: Number of Participants Who Completed the PCORI Ways of Engaging-Engagement Activity Tool (WE-ENACT) Patient and Stakeholder Survey
Description: The investigators will measure engagement from the community partner perspective using the PCORI WE-ENACT Patient and Stakeholder Survey, completed annually. This measure includes items to describe engagement from the stakeholder's point of view. One or two key representatives from each community partner agency will participate.
  The Outcome Measure Data Table includes the number of participants who completed the survey.
Time Frame: Baseline and every 12 months assessed up to month 48.
Measure: Count of Participants; unit: Participants
Groups:
- Stakeholders: Partners for the proposed research include representatives from the community agencies already engaged in developing the current proposal, including local government agencies, CBOs that serve Veterans, and VSOs; an individual Veteran with DM with experience and expertise in use of VHA and community resources; the MEDVAMC DM educator; and leadership from the VHA research team. These community-VHA partners will meet twice a year in person or online during the project to discuss progress and study updates and provide input on key aspects of study implementation, data collection and analysis, and dissemination of findings. Specific topics for each meeting will depend on the stage of the study at the time of the meeting. Potential topics include troubleshooting problems with participant recruitment or retention; addressing challenges encountered by peer mentors; discussion and interpretation of study outcomes; and opportunities for dissemination of findings to key community, government, and VHA stakeholders. All members of the partnership who are not VHA employees will be compensated $150 per meeting in recognition of their time and expertise.
Arm/Group | Stakeholders
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were captured from informed consent through the last follow-up assessment (Month 6) or participant withdrawal.
Description: The following types of events were considered adverse events (AEs) for this minimal-risk study. No other AEs were captured. Specific AE terms were not captured.
  1. Marked deterioration in depressed or anxious mood
  2. Development of manic or psychotic symptoms
  3. Suicidal and homicidal ideation
  4. Suicide attempt
  5. Incident of violence toward others
  6. Hospitalization for acute medical or psychological illness
  7. Any other life-threatening or potentially disabling event
  8. Death
Arm/Group | iNSPiRED | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/110 | 0/108
Serious Adverse Events (participants affected / at risk) | 12/110 | 11/108
Other Adverse Events (participants affected / at risk) | 1/110 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNSPiRED (N=110) | Usual Care (N=108)
Hospitalization (Vascular disorders) | 3 (3) | 1 (1)
Death (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hospitalization (Cardiac disorders) | 2 (2) | 3 (4)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hospitalization (General disorders) | 3 (3) | 0 (0)
Hospitalization (Psychiatric disorders) | 2 (2) | 0 (0)
Hospitalization (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hospitalization (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iNSPiRED (N=110) | Usual Care (N=108)
Homicidal ideation (Social circumstances) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Connecting participants to medical care and resources for diabetes and mental health self-management was a primary component of the peer coaching intervention. The COVID-19 pandemic reduced the availability of these resources. The impact of reduced availability of resources on the study results is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04041375/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04041375/ICF_002.pdf